CLINICAL TRIAL: NCT01503593
Title: Phase 3 Study of Using Combination of Bi Phasic Calcium Phosphate and Bu Phasic Calcium Sulphate During Extractions
Brief Title: Using Combination of Synthetic Bone Substitutes During Extractions
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0326-11-RMB; 0362-11-RMB
Record Dates: First submitted 2011-12-18; First posted 2012-01-04 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Periodontitis; Dental Caries; Alveolar Bone Losses
MeSH Terms: conditions — Periodontitis; Dental Caries; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alveolar ridge dimensions (No Intervention): Control group - Only extraction teeth
- Alverolar ridge dimension (Experimental): Extraction of teeth and implant a bone substitute
  Interventions: Device: Calcium Phosphate, Calcium Sulphate

INTERVENTIONS:
Device: Calcium Phosphate, Calcium Sulphate — 1cc of Calcium Phosphate and 1cc of Calcium Sulphate
  Arms: Alverolar ridge dimension

SUMMARY:
The study was designed to assess the effectiveness of conservation ridge preservation (horizontal and vertical dimension) after tooth extraction with and without combination of bone substitutes based on synthetic (calcium sulfate mixed with phosphate.

DETAILED DESCRIPTION:
Using the combination of these two bone substitute is taken in order to diminish the alveolar ridge alternations after tooth extraction. the investigator will measure the horizontal and vertical changes (primary outcome) and the adverse effects (secondary outcome)in 4 months period

ELIGIBILITY:
Inclusion Criteria:

1. Patients over age 18.
2. Patients who require extraction of teeth for Periodontal or other dental reasons (up one tooth in each quarter when there are existing adjacent teeth).

Exclusion Criteria:

1. Inability to pass informed consent procedure
2. Pregnant women
3. Breastfeeding women
4. Patient taking medications that affect bone metabolism such as bisphosphonates
5. Extractions sites contaminated
6. Smoking over 10 cigarettes a day
7. Patients with removable prostheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
The change of the dimension of the alveolar ridge | Immediatly after tooth extraction (up to 10 minutes after the extraction) and 4 monthes after extraction
  Measurement of socket width (aspect B/L) at three points Height:
  1. Record-high ridge (buccal/lingual-palatal )
  2. 3 mm apically to the peak ridge (buccal/lingual-palatal )
  3. 6mm apically to the peak ridge (buccal/lingual-palatal )
  Measurement of alveolar ridge height:
  Measured distance between the summit crater and the peak of the ridge and the center line connecting the CEJ of adjacent teeth

SECONDARY OUTCOMES:
Post operative adverse effects | immediate after the extraction and until 4 monthes after
  The investigators will record the optionally adverse effect such as edema, infection, pain, exposure of the membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Mayer, D.M.D., Principal Investigator — Rambam Health Care Campus, Haifa, Israel